CLINICAL TRIAL: NCT01912755
Title: Anesthetic Efficacy of 4% Articaine (Mandibular Infiltration) and 2% Lidocaine (Alveolar Nerve Block), Associated With 1:100.000 Epinephrine, in Lower Molars With Irreversible Pulpits
Brief Title: Anesthetic Efficacy of Articaine and Lidocaine in Lower Molars With Irreversible Pulpits
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Francisco Groppo, Professor of Physiological Sciences Department, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-10834-4
Record Dates: First submitted 2013-07-19; First posted 2013-07-31 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Irreversible Pulpitis; Pain
Keywords: Pulpitis; Hot tooth; Articaine; Lidocaine; Local anesthetics
MeSH Terms: conditions — Pain; Pulpitis | interventions — Carticaine; Epinephrine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Articaine (Experimental): injection of 1.8 mL buccal infiltrations of 4% articaine with 1:100,000 epinephrine in one tooth with a clinical diagnosis of symptomatic irreversible pulpitis.
  Interventions: Drug: 4% articaine with 1:100,000 epinephrine; Drug: 2% lidocaine with 1:100,000 epinephrine
- Lidocaine (Active Comparator): 1.8 mL 2% lidocaine with 1:100,000 epinephrine injected as inferior alveolar nerve block in the mandible side with one tooth with a clinical diagnosis of symptomatic irreversible pulpitis.
  Interventions: Drug: 4% articaine with 1:100,000 epinephrine; Drug: 2% lidocaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: 4% articaine with 1:100,000 epinephrine — If the primary anesthesia failed after ten minutes, an intraligamentary injection with 4% articaine with 1:100,000 epinephrine was performed and the procedure initiated. When access to the pulp chamber was available, intrapulpal anesthesia was given using 4% articaine with 1:100,000 epinephrine.
  Other Names: articaine
Drug: 2% lidocaine with 1:100,000 epinephrine — If the patient reported pain during treatment and access to the pulp chamber was not achieved, an IANB was performed with 2% lidocaine with 1:100,000 epinephrine.
  Other Names: Lidocaine

SUMMARY:
The aim of this study was to verify the effectiveness of an anesthetic called articaine for dental treatment, comparing it with an anesthetic commonly used in dental clinic: lidocaine. Two types of local anesthesia (oral injection) in accordance with the solution used were performed. For patients anesthetized with articaine, an injection of anesthesia close to the tooth to be treated was used. For the anesthetic lidocaine an injection on the cheek at the bottom of the mouth was made. Differences between both techniques are mainly regarding the area of numbness. In the injection with articaine only a small part of the lip and the tooth was anesthetized. With lidocaine injection, the lower region of the entire side of the tooth and half of the tongue on the same side was numbed. The treatment was electronic randomized and there was equal chance to one or another treatment. The investigators are studying this new form of anesthesia (near the tooth that was treated) to see if it can numb the tooth to an emergency treatment, if it really decreases the feeling of numbness and discomfort during the service. Patients receiving articaine were submitted to cone beam exam at no cost.

DETAILED DESCRIPTION:
Aim: This randomized clinical trial compared the anesthetic efficacy of buccal infiltration (BI) with 4% articaine (AR) and inferior alveolar nerve block (IANB) with 2% lidocaine (LI), both with 1:100,000 epinephrine, in symptomatic mandibular molars with irreversible pulpitis. Likewise, we compared the efficacy of the primary infiltration (BI or IANB) with one supplemental injection (intraligamentary infiltration with articaine for AR and BI with articaine for LI). The influences of buccal cortical bone thickness and root distances to buccal cortical bone on articaine performance (AR) were also evaluated using cone-beam tomography. methodology: Volunteers presenting symptomatic mandibular molars with irreversible pulpitis were randomly divided into two groups (30 for AR and 20 for LI). Success was recorded when complete pain-free treatment was achieved after primary injection or when one supplemental injection was needed for emergency endodontic procedures.

ELIGIBILITY:
Inclusion Criteria:

* long-lasting moderate to severe pain during cold test
* absence of periapical radiolucency except for a widened periodontal ligament (evaluated in periapical radiographs)
* vital coronal pulp on access opening

Exclusion Criteria:

* Previous history of allergy to local anesthetics
* Subjects with systemic diseases
* Pregnancy and lactation
* Subjects taking any kind of medication that could change or influence the outcome of this research
* Subjects without painful symptoms
* Negative thermal testing, periapical lesion, incomplete root formation, presence of fistula or abscess, cracks or fractures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pain perception 3 | 10 minutes after injection
  Patients received visual analogue scales (VAS) to record their pain perception ten minutes after local anesthetic injection.

SECONDARY OUTCOMES:
Buccal cortical bone thickness | one week after injection
  Cone-beam computed tomography scans (iCat, Imaging Science, USA) were taken from patients submitted to articaine injection in order to measure the buccal cortical bone thickness.
Root distance to the bone | one week after injection
  Cone-beam computed tomography scans (iCat, Imaging Science, USA) were taken from patients submitted to articaine injection in order to measure the the distance between the mesial and lingual roots to the buccal cortical bone.
Basal pain perception | 10 minutes before injection
  Patients received visual analogue scales (VAS) to record their pain perception 10 min before the local anesthetic injection.
Pain perception 2 | 5 minutes before injection
  Patients received visual analogue scales (VAS) to record their pain perception 5 min before the local anesthetic injection (after the cold testing).

CONTACTS AND LOCATIONS:
Overall Officials: José FA Almeida, DDS, PhD, Study Chair — Endodontics Area - FOP-UNICAMP; Maria RF Monteiro, DDS, MSc, Principal Investigator — Endodontics Area - FOP-UNICAMP
Locations (1):
- Piracicaba Dental School - UNICAMP, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Aggarwal V, Jain A, Kabi D. Anesthetic efficacy of supplemental buccal and lingual infiltrations of articaine and lidocaine after an inferior alveolar nerve block in patients with irreversible pulpitis. J Endod. 2009 Jul;35(7):925-9. doi: 10.1016/j.joen.2009.04.012. PMID 19567309
- [Background] Ashraf H, Kazem M, Dianat O, Noghrehkar F. Efficacy of articaine versus lidocaine in block and infiltration anesthesia administered in teeth with irreversible pulpitis: a prospective, randomized, double-blind study. J Endod. 2013 Jan;39(1):6-10. doi: 10.1016/j.joen.2012.10.012. Epub 2012 Nov 13. PMID 23228249
- [Background] Berlin J, Nusstein J, Reader A, Beck M, Weaver J. Efficacy of articaine and lidocaine in a primary intraligamentary injection administered with a computer-controlled local anesthetic delivery system. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Mar;99(3):361-6. doi: 10.1016/j.tripleo.2004.11.009. PMID 15716846
- [Derived] Monteiro MR, Groppo FC, Haiter-Neto F, Volpato MC, Almeida JF. 4% articaine buccal infiltration versus 2% lidocaine inferior alveolar nerve block for emergency root canal treatment in mandibular molars with irreversible pulpits: a randomized clinical study. Int Endod J. 2015 Feb;48(2):145-52. doi: 10.1111/iej.12293. Epub 2014 May 22. PMID 24702239